CLINICAL TRIAL: NCT02724917
Title: A Phase 1b/2a, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of APN1125 in Subjects With Schizophrenia
Brief Title: Safety, Tolerability, and Pharmacokinetics of APN1125 in Subjects With Schizophrenia
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted by sponsor for business reasons
Sponsor: CoMentis (Industry)
Collaborators: Alpharmagen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN1125-002
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- APN1125, Low Dose (Experimental): APN1125, Low Dose
  Interventions: Drug: APN1125
- APN1125, Mid Dose (Experimental): APN1125, Mid Dose
  Interventions: Drug: APN1125
- APN1125, High Dose (Experimental): APN1125, High Dose
  Interventions: Drug: APN1125
- Placebo (Placebo Comparator): Placebo to match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APN1125 — Oral solid dose form of APN1125
  Arms: APN1125, High Dose; APN1125, Low Dose; APN1125, Mid Dose
Drug: Placebo — Placebo to match
  Other Names: Placebo to match
  Arms: Placebo

SUMMARY:
The purpose of this study in patients with schizophrenia is to evaluate the safety, tolerability, and pharmacokinetics of 3 doses (low, mid, high) of APN1125 compared with placebo when administered as repeated daily oral doses.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety profile, tolerability and pharmacokinetics (PK) of APN1125 following 14 days of once-daily oral dosing in subjects with schizophrenia on stable second-generation antipsychotic therapy.

This is a randomized, double-blind, 2-week, multiple ascending dose study of APN1125. This study will enroll up to three sequential cohorts of subjects diagnosed with schizophrenia, each randomly assigned to receive one of three doses (low, medium, or high) of APN1125 or matching placebo. Following admission to an Early Phase Clinical Unit (EPCU), APN1125 will be administered once daily for 2 weeks. All subjects will remain confined to the EPCU for a total of 20 days, consisting of admission, dosing and observation periods.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race
* 18 to 45 years of age, inclusive
* Diagnosed with schizophrenia, as defined in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), in a non-acute (e.g., chronic) phase and clinically stable for at least 12 weeks before screening
* Currently on a stable second-generation anti-psychotic regimen (stable dose and medication for 12 weeks)
* Subjects (male and female) of childbearing potential must use two effective methods of contraception starting from the time of providing informed consent throughout the duration of the study and for 3 months after discharge
* Women of childbearing potential must have a negative pregnancy test at screening and at admission

Exclusion Criteria:

* Clinically significant abnormal serum electrolytes (sodium, potassium, calcium, and magnesium) after repeat testing
* Insulin-dependent diabetes or insufficiently controlled diabetes mellitus in the judgment of the Investigator
* Renal insufficiency with serum creatinine >1.6 mg/dL Malignant tumor within the 5 years before Screening with the exception of treated squamous and basal cell carcinoma, cervical carcinoma in situ, or brachytherapy for localized prostate cancer
* Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
* Unstable medical condition that is clinically significant in the judgment of the Investigator
* Body mass index (BMI) >38 kg/m^2 at Screening ALT or AST >1.5 times the upper limit of normal
* Positive serology for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 and/or 2 antibodies
* Untreated clinically significant hypo- or hyperthyroidism; treated hypo- or hyperthyroidism should be stable for at least 8 weeks prior to Screening
* History of myocardial infarction or unstable angina within 6 months before Screening
* Cardiovascular disease history including symptomatic hypotension (supine systolic blood pressure [SBP] <90 mmHg or supine diastolic blood pressure [DBP] <60 mmHg), symptomatic orthostatic hypotension (orthostatic change in SBP >20 mmHg or DBP >15 mmHg), or hypertension (supine SBP >160 mmHg or supine DBP >95 mmHg ) or significant cardiac arrhythmia (in the judgment of the Investigator)
* Clinically significant abnormality on Screening or Baseline electrocardiogram (ECG), including but not necessarily limited to a confirmed QTcF (QT interval corrected for heart rate using Fridericia's formula) interval value >450 msec for males or >470 msec for females
* Current treatment with more than 2 atypical antipsychotics Psychiatric hospitalization due to breakthrough psychotic symptoms or acute exacerbations within 3 months before Day -1. Subjects with a recent "social" hospitalization may be screened after consultation with the Medical Monitor.
* Subjects with other DSM-5 disorders are ineligible if the comorbid condition is clinically unstable or has been the primary focus of treatment within 3 months prior to Screening
* Subjects meeting DSM-5 criteria for moderate to severe alcohol or substance use disorder (other than nicotine- or caffeine-related disorders) within 6 months prior to Screening
* Urine drug screen (UDS) positive for drugs of abuse (excluding prescribed benzodiazepines) or positive alcohol breath test at Screening and/or Baseline (may be repeated once if, in the judgment of the Investigator, the subject does not meet DSM-5 criteria for moderate to severe substance abuse disorder)
* Significant suicide risk as defined by 1) suicidal ideations as endorsed on items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the year prior to Screening or Baseline, 2) suicidal behaviors within the 2 years prior to Screening, or 3) Investigator assessment
* History of stroke, brain tumor, subdural hematoma, Parkinson's Disease, dementia or other clinically significant neurological condition
* Head trauma with loss of consciousness within 12 months prior to Screening
* Active acute or chronic CNS infection
* History of a seizure disorder
* Immunosuppressants, including systemic corticosteroids (administered at an immunosuppressant dose in the judgment of the Investigator) (Note: Inhaled, nasal, or topical steroid use for allergy or other inflammation is permitted)
* Any drugs with CNS activity (Note: Occasional (as needed) use of a sedative-hypnotic (e.g., benzodiazepine or nonbenzodiazepine [e.g., zolpidem, zaleplon, zopiclone, and eszopiclone]) as a sleep aid and stable second generation psychotics are permitted)
* Prohibited antipsychotic medications (e.g., clozapine or typical, first-generation antipsychotics)
* Excessive alcohol consumption (regular alcohol intake 14 units per week or more) or has a history of alcohol use disorder. Use of alcohol up to 48 hours before admission to the EPCU is not allowed.
* Failure or inability to perform Screening or Baseline assessments
* Exposure to an experimental drug or experimental medical device within 2 months before Screening, or an experimental biologic within 3 months before Screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of APN1125 in subjects with schizophrenia via adverse events | 25 days
Assessment of safety and tolerability of APN1125 in subjects with schizophrenia via vital signs (e.g., blood pressure, pulse rate, respiratory rate, oral temperature) | 25 days
Assessment of safety and tolerability of APN1125 in subjects with schizophrenia via ECGs | 25 days
Assessment of safety and tolerability of APN1125 in subjects with schizophrenia via physical exams | 25 days
Assessment of safety and tolerability of APN1125 in subjects with schizophrenia via clinical laboratory tests (chemistry, hematology, coagulation and urinalysis) | 25 days

SECONDARY OUTCOMES:
Maximum observed plasma APN1125 concentration (Cmax) | Days 1 and 14
Time corresponding to occurrence of Cmax (Tmax) | Days 1 and 14
Area under the Curve from time zero to the last quantifiable plasma APN1125 concentration (AUClast) | Days 1 and 14
Area under the Curve from time zero extrapolated to plasma APN1125 concentration at infinity (AUCinf) | Days 1 and 14
Terminal plasma APN1125 rate constant (lambda z) | Days 1 and 14
Apparent plasma APN1125 terminal half-life (t1/2) | Days 1 and 14
Apparent APN1125 plasma clearance (CL/F) | Days 1 and 14
Amount of unmetabolized APN1125 excreted in urine (Ae) | Days 1 and 14
Fraction of unmetabolized APN1125 dose excreted in urine (Fe) | Days 1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: David P Walling, PhD, Principal Investigator — Collaborative Neuroscience Network
Locations (1):
- Collaborative Neuroscience Network, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No